CLINICAL TRIAL: NCT06078059
Title: Mechanisms of Treatment Effects Using Cultured, Allogeneic Mesenchymal Stromal Stem Cells (MSCs) in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Blood Transfusion Centre of Slovenia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMC Ljubljana
Record Dates: First submitted 2023-07-23; First posted 2023-10-11 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee; Osteoarthritis; Mesenchymal stem cells; Allogeneic
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Knee aspiration and the application of UCB-MSCs
  Interventions: Biological: Knee aspiration + UCB-MSCs
- Control group (Active Comparator): Only knee aspiration, without the application of UCB-MSCs
  Interventions: Other: Knee aspiration

INTERVENTIONS:
Biological: Knee aspiration + UCB-MSCs — Knee aspiration and the application of cultered allogeneic umbilical cord blood-derived mesenchymal stromal stem cells (UCB-MSCs).
  Arms: Intervention group
Other: Knee aspiration — Knee aspiration
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to pharmacologically evaluate the effects of culturued allogeneic umbilical cord blood-derived mesenchymal stromal stem cell (UCB-MSCs) in the treatment of end-stage knee osteoarthritis (Kellgren-Lawrence grade 4) with the analysis of soluble biomarkers and expression of key genes, as well as the evaluation of clinical outcomes with patient-reported outcome measures (PROMs) and recording of potential complications.

Patients will be randomized in the intervention and control groups. In both groups, the knee aspiration will be performed 4-6 weeks prior to the knee arthroplasty to analyse baseline synovial fluid characteristics. The intervention group will receive the injection of UCB-MSCs. All patients will complete PROMs questionnaires and maintain a pain diary on visual analogue scale (VAS) at home until the surgery. On the day of admission to hospital for knee arthroplasty, the same questionnaires will be administered again. During the operative procedures, the samples of synovial fluid, synovial membrane and resected cartilage will be obtained and analysed afterwards.

It is anticipated that the study results will contribute to elucidate the mechanisms of action of MSCs in the treatment of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage (Kellgren-Lawrence) knee osteoarthritis scheduled for knee arthroplasty
* Osteoarthritis of primary or post-traumatic etiology

Exclusion Criteria:

* Secondary arthritis of other etiology
* Rheumatic diseases
* Uncontrolled metabolic disorders
* Crystalopathies
* Coagulopathy
* Anticoagulant therapy
* Heart failure
* Renal failure
* Other conditions that may affect immune response or pose additional risk during cell application

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Soluble biomarkers analysis with multiplex bead-based immunoassays Luminex in synovial fluid | After sampling
  Luminex assay is a type of immunoassay that precisely measures multiple analytes in one sample. It is a bead-based immunoassay that allows for multiplex detection of analytes simultaneously. Color-coded microspheres or beads are internally dyed with different proportions of red and infrared fluorophores that correspond to a distinct spectral signature or bead region. The quantification of multiple cytokines and other biomarkers in samples provides critical information about biological processes and diseases.
Biomarkers analysis with Enzyme-linked immunosorbent assay (ELISA) in synovial fluid | After sampling
  Enzyme-linked immunosorbent assay (ELISA) is the main approach for the sensitive quantification of protein biomarkers in body fluids and is currently employed in clinical laboratories for the measurement of clinical markers. It also constitutes the main methodological approach for biomarker validation and further qualification.
Quantitative real-time PCR (qRT-PCR) analysis of gene expression in chondrocytes and synoviocytes | After sampling
  Quantitative real-time PCR (qRT-PCR) is a major development of PCR technology that enables reliable detection and measurement of products generated during each cycle of PCR process. The detection of changes in fluorescence intensity during the reaction enables to follow the PCR reaction in real time. qRT-PCR is comprised of several steps: 1. RNA is isolated from target tissue/cells, 2. mRNA is reverse-transcribed to cDNA, 3. modified gene-specific PCR primers are used to amplify a segment of the cDNA of interest, following the reaction in real time, 4. the initial concentration of the selected transcript in a specific tissue or cell type is calculated from the exponential phase of the reaction.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 4-6 prior to surgery and at admission
  Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Pain on Visual Analogue Scale (VAS) | 4-6 prior to surgery and at admission
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('the worst pain imaginable').
EuroQol 5-Dimensions 3-Levels (EQ-5D-3L) questionnaire | 4-6 prior to surgery and at admission
  EQ-5D-3L descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression . Each dimension has 3 levels: no problems, some problems, and extreme problems. The respondent is asked to indicate his or her health state by ticking the box that marks the most appropriate level of problems in each dimension. A unique health state can be described according to the responses to the 5 questions. Health states defined in this way may be converted into a single summary index by applying a formula that attaches values to each of the levels in each dimension. States can be converted to a single value where 1 is equivalent to full health and 0 to a state equivalent to death.
EuroQol self-rated health on Visual Analogue Scale (EQ-VAS) | 4-6 prior to surgery and at admission
  EQ-VAS records the patient's self-rated health on a vertical visual analogue scale from 0 to 100, where 0 represents the worst health state imaginable and 100 represents the best health state imaginable.
Serious Adverse Events (SAE) | Until 1 month after the application of UCB-MSCs
  Serious adverse events (SAE) are defined as any complication requiring hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Matej Drobnič, MD, PhD, Principal Investigator — University Medical Centre Ljubljana; Urban Švajger, MPharm, PhD, Principal Investigator — Blood Transfusion Centre of Slovenia
Locations (1):
- University medical centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svajger U, Kolar M, Kobold A, Drobnic M. Mechanisms of treatment effects using allogeneic, umbilical cord-derived mesenchymal stromal stem cells (MSCs) in knee osteoarthritis: a pharmacological clinical study protocol. Trials. 2024 Aug 13;25(1):533. doi: 10.1186/s13063-024-08360-x. PMID 39135209